CLINICAL TRIAL: NCT00241995
Title: Antiglutamate Anticonvulsants in the Treatment of Alcohol Withdrawal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-RCT_LOND_GAT_AWS_2003
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-10

CONDITIONS: Topiramate; Lamotrigine; Memnatine; Diazepam; Placebo
MeSH Terms: interventions — Anticonvulsants

INTERVENTIONS:
Drug: Anticonvulsants

SUMMARY:
The study is aimed to evaluate the efficacy of antiglutamate anticonvulsants (topiramate, lamotrigine, and memantine) in the treatment of alcohol withdrawal syndrome

ELIGIBILITY:
Inclusion Criteria:

Alcohol dependence Alcohol withdrawal syndrome

Exclusion Criteria:

Drug dependence Major psychiatric diagnoses Severe somatic illness

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny M Krupitsky, MD, PhD, Principal Investigator — St. Petersburg State Pavlov Medical University